CLINICAL TRIAL: NCT06378411
Title: Development and Application of a Musical Game for Motor Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade da Madeira (Other)
Responsible Party: Principal Investigator, Yasmim Fernandes Moniz, Master in Biomedical Engineering, Universidade da Madeira
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: P109
Record Dates: First submitted 2024-04-18; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Health People; Survivors of Stroke
Keywords: music intervention; rehabilitation; stroke; motor coordination; adults
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music Game Group (Experimental): Use of Moniz Game with digital interface
  Interventions: Device: Music Game Intervention
- Music Game Controller Group (Experimental): Use of Moniz Game with piano controller
  Interventions: Device: Music Game Intervention
- Music Practice Group (Active Comparator): Use of music trainning as intervention
  Interventions: Device: Music Game Intervention

INTERVENTIONS:
Device: Music Game Intervention — Use of music to induce improvements in cognitive and motor outcomes.
  Other Names: Music Based Intervention

SUMMARY:
The aim of this study is to develop, adapt a musical game for residents of RAM, and evaluated the usability and correlation between this game with the improvement of motor coordination in short time.

ELIGIBILITY:
Inclusion Criteria:

* Health people
* Survivors of Stroke

Exclusion Criteria:

* Dementia
* Visual Defict
* People who already knows how to play piano

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Motor Coordination | 1 month
  Motor Performance by time
Usability | 20 minutes
  Evaluated the quality with the facility to use the system

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade da Madeira, Funchal, Portugal

IPD SHARING:
Plan to Share IPD: No